CLINICAL TRIAL: NCT03832296
Title: Independent Weight Loss Maintenance for Communities With Arthritis in North Carolina: the I-CAN Clinical Trial
Acronym: I-CAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00033618.I-CAN
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2020-11

CONDITIONS: Osteo Arthritis Knee
Keywords: Arthritis; Knee; weight loss
MeSH Terms: conditions — Arthritis; Weight Loss

STUDY DESIGN:
Intervention Model Description: Participants will include 212 older adults aged ≥ 51 yrs. with knee OA who achieved a weight loss ≥ 5% in the D+E intervention arm of the WE-CAN trial. Eligible WE-CAN D+E participants will be randomized to either the weight-loss maintenance or health education attention control groups.
Who Masked: Outcomes Assessor
Masking Description: Each eligible participant will be randomized to one of the two arms of the clinical trial (weight-loss maintenance, control) according to a variable block-length algorithm that will be controlled by the Data Management Group. Randomization will be stratified by intervention site to ensure nearly equal sample sizes for the two interventions to balance local population characteristics. Randomization uses a web-based system that is part of the study data management system. Intervention visits will not include any assessments and outcome assessors will remain blinded to group assignment. The lead biostatistician of the Data Management Group will develop the randomization table.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight-Loss Maintenance (Experimental): Weight Loss Maintenance Intervention
  Interventions: Behavioral: Weight-Loss Maintenance
- Health Education (Attention Control) (Active Comparator): Health Education Intervention
  Interventions: Behavioral: Health Education (Attention Control)

INTERVENTIONS:
Behavioral: Weight-Loss Maintenance — Over the course of the first 6-months, participants will build their self-efficacy to maintain weight loss on their own, empowered to do what is needed to achieve personal goals and long-term behavior change (months 7-18). The first 6 months of I-CAN will prepare participants for successful independent weight-loss maintenance in months 7-18. During the 12-month independent weight-loss maintenance phase participants exercise on their own and maintain their weight loss (or increase weight loss if they choose) with the only contact from interventionists being two newsletters at months 9 and 15.
  Arms: Weight-Loss Maintenance
Behavioral: Health Education (Attention Control) — Participants in the control group will attend an individual session during month 1, and a monthly face-to-face group meeting during months 2-6. The sessions will provide attention, social interaction, and physician-based health education. Participants will receive a newsletter during months 9 and 15.
  Arms: Health Education (Attention Control)

SUMMARY:
The study team is currently conducting a pragmatic, community-based assessor-blinded randomized controlled trial (RCT) in overweight and obese adults > 50 years with knee OA in both urban and rural counties in North Carolina. As the participants randomized to the 18 month diet and exercise group in the WE-CAN study successfully complete the intervention (≥ 5% weight loss), the study team has the unique opportunity to evaluate the effectiveness of a theoretically-based tapered weight maintenance intervention. Eligible participants will be randomized to either the weight-loss maintenance or health education attention control groups.

DETAILED DESCRIPTION:
Results from the Intensive Diet and Exercise for Arthritis (IDEA) trial showed that 10% diet-induced weight loss combined with exercise (D+E) was twice as effective at relieving knee pain and improving function and mobility as previous long-term weight loss and exercise programs in similar cohorts. The treatment effects of D+E on these clinical outcomes were mediated by changes in self-efficacy over the course of the trial. However, most people tend to regain most or all of the lost weight in three to five years. The challenge is maintaining the weight loss and sustaining the efficacy of the intervention.

Our current trial (WE-CAN) is designed to adapt the successful IDEA intervention to real-world clinical and community settings. As WE-CAN participants in the D+E group complete their intervention, the investigators will leverage our organizational infrastructure to maintain weight-loss without supervised intervention by increasing participant confidence to establish and adhere to a routine of good exercise and diet behaviors independently.

Participants will include 212 older adults aged ≥ 51 yrs. with knee osteoarthritis (OA) who achieved a weight loss ≥ 5% in the D+E intervention arm of the WE-CAN trial. All WE-CAN participants meet the ACR clinical criteria for knee OA, which includes knee pain on most days of the week plus at least three of the following six: age ≥ 50 years, stiffness < 30 min/day, crepitus, bony tenderness, bony enlargement, and/or no palpable warmth. Eligible WE-CAN D+E participants will be randomized to either 6-month facilitated weight-loss maintenance or health education control interventions. The primary aim is to compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on maintaining weight loss subsequent to a 12-month unsupervised follow-up period. Secondary aims will compare the two interventions on WOMAC knee pain and function, health-related quality of life (SF-36), 6-minute walk distance, and weight-loss maintenance self-efficacy following the 12-month unsupervised period. The study team will also establish the cost-effectiveness of a 6-month facilitated weight-loss maintenance intervention for older adults with knee OA by conducting cost-effectiveness and budgetary impact analyses using data from the current trial in a validated computer-simulated model of knee OA.

There have been numerous attempts to prevent weight regain in adults. This study is significant in that it is designed to encourage older adults with knee OA that have experienced significant weight loss to develop strategies that will build self-efficacy for maintaining weight loss on their own long after the active intervention ends.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 51
* achieved a weight loss ≥ 5% in the D+E intervention arm of the WE-CAN trial

Exclusion Criteria:

* Weight loss < 5% of baseline body weight
* Significant co-morbid disease that would threaten safety or impair ability to participate in interventions or testing (Blindness; Type 1 diabetes; Severe coronary artery disease)
* Inability to finish 18-month study or unlikely to be compliant (Planning to leave area > 2 month during the next 18 months)

Min Age: 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Weight-Loss Maintenance | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on maintaining weight loss subsequent to a 12-month unsupervised follow-up period.

SECONDARY OUTCOMES:
Knee Pain measured by the WOMAC Index | 18 Months
  The investigators will measure self-reported pain using the WOMAC (scores will be pulled from the KOOS Questionnaire in which the WOMAC is embedded). The pain index assesses participants' pain on a scale, ranging from 0 (none) to 4 (extreme). The pain subscale consists of 5 items and total scores can range from 0-20, with larger scores indicating greater dysfunction.
Function measured by the WOMAC Index | 18 Months
  The investigators will measure self-reported physical function using the WOMAC (scores will be pulled from the KOOS Questionnaire in which the WOMAC is embedded). The LK version asks participants to indicate on a scale from 0 (none) to 4 (extreme) the degree of difficulty experienced in the last week due to knee OA. Individual scores for the 17 items are totaled to generate a summary score that could range from 0-68, with higher scores indicating poorer function.
Health Related Quality of Life: SF-36 | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on health-related quality of life (SF-36) subsequent to a 12-month unsupervised follow-up period. Two summary scores are acquired: physical health and mental health. Range=0-100. Higher scores indicate better health.
Mobility- 6 minute walk test | 18 Months
  The primary mobility measure will be 6-minute walk distance. Participants are told to walk as far as possible in 6 minutes on an established course.
Self-Efficacy - Perceived Stress: questionnaire | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on self-efficacy. The perceived stress questionnaire will measure the degree to which people perceive their lives as stressful. Range = 0-40. Higher numbers indicate higher stress.
Self-Efficacy - Walking Efficacy for Duration: walking efficacy for duration scale | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on self-efficacy. The walking efficacy for duration scale measures one's ability to walk/jog at a moderately fast pace for various durations. Range 0-100. A higher score indicates a higher self-efficacy.
Self-Efficacy - PANAS | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on self-efficacy. The Positive and Negative Affect (PANAS) measures both positive and negative affect, leading to more insightful outlooks regarding participants' feeling states. This scale consists of 20 items that reflect the intensity of how the participant "feels" right now. Range=10-50 for each subscale. A higher score for positive affect indicates a higher level of positive affect. A higher score for negative affect indicates a higher level of negative affect.
Self-Efficacy - Gait Efficacy - gait efficacy/environmental efficacy scale | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on self-efficacy. The gait efficacy/environmental efficacy scale will ask the participants' confidence in performing certain activities. Confidence in performing activities. Participants will be asked to indicate their level of confidence being able to complete different tasks. Range=0-100. A higher score indicates higher self-efficacy.
Self-Efficacy - Satisfaction with Life: Satisfaction with life scale | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on self-efficacy. The Satisfaction with life scale is focused to assess global life satisfaction. Range=5 to 35. A higher scale indicates a higher level of life satisfaction.
Self-Efficacy - Weight Efficacy Scale | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on self-efficacy. The Weight Efficacy Lifestyle Questionnaire (WEL) is a 20-item measure employed to assess self-efficacy for weight management. Range=0 to 180. Higher numbers indicate better confidence.
Self-Efficacy - Adherence Self Efficacy Scale | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on self-efficacy. The adherence questionnaire is designed to assess beliefs in one's ability (confidence) to continue exercising at various intensities and frequencies. Range=0-100. A higher score indicates higher self-efficacy.
Self-Efficacy - Barriers Self-Efficacy to Exercise | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on self-efficacy. The Barriers Self-Efficacy to Exercise measures confidence in dealing with barriers to exercise. Range=0-100. Higher numbers indicate higher confidence.
Self-Efficacy - Multidimensional Outcome Expectations for Exercise Scale (MOEES): questionnaire | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on self-efficacy. The MOEES questionnaire consists of three subscales: physical outcome expectations (score range 6-30), social outcome expectations (score range 4-20), and self-evaluative outcome expectations (score range 5-25). Each subscale is scored by summing the numerical ratings for each response. Higher scores are indicative of higher levels of outcome expectations for exercise.
Self-Efficacy - Perceived Barriers: questionnaire | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on self-efficacy. The perceived barriers questionnaire measures a person's perceptions to barriers to performing exercise. The questionnaire is scored by finding the mean for each response (range = 1-5). Higher scores indicate higher perception of barriers.
Self-Efficacy - Weight Loss Maintenance: questionnaire | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on self-efficacy for maintaining weight loss. Range=0-100. Higher scores indicate more confidence in maintaining weight loss.
Cost-Effectiveness | 18 Months
  Resource utilization will be collected by questionnaire. MD and non-MD office visits will be collected via self-report with domains including visits to clinicians (physicians, nurses, physical therapists, others), tests, medications, injections, surgery, alternative therapies. The number of visits associated with utilization of each of 4 domains, MD visits, non-MD visits, ED visits, and inpatient stays, will be examined.
Cost-Effectiveness- WPAI | 18 Months
  The Work Productivity and Activity Impairment index (WPAI) will be used to assess absenteeism and reduced productivity while at work (presenteeism). Outcome (OC) scores can be derived from the WPAI: OC1, percent work time missed due to health, (percentage of absenteeism); percent impairment while working due to health, (percentage of presenteeism); percent overall work impairment due to health, percent activity impairment due to health. For all 4 outcomes, greater scores (range 0-100%) indicate greater impact of health.

OTHER OUTCOMES:
Mobility - SPPB & GaitRite | 18 Months
  The Short Physical Performance Battery (SPPB) will be used to measure mobility. The SPPB is comprised of the following tests (balance, walking speed, and chair rise). The scores range from 0 (worst performance) to 12 (best performance). Mobility will also be measured using the GaitRite.
Mobility - stair activity | 18 Months
  A test of ascending and descending stair activity measured by the time (in seconds) it takes to ascend and descend a flight of 8 steps with 20cm (8 inch) step height and handrail will also be performed.
Pain Catastrophizing Scale (PCS) | 18 Months
  The PCS questionnaire will be used to assess catastrophizing (rumination, magnification, and helplessness). The PCS total score is computed by summing responses to all 13 items. PCS total scores range from 0 - 52. Lower scores indicate less pain.
Knee injury and Osteoarthritis Outcome Score (KOOS) | 18 Months
  The KOOS questionnaire will be used to assess the patient's opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury and also consequences of primary osteoarthritis (OA). It holds 42 items in five separately scored subscales: 1) KOOS Pain; (2) KOOS Symptoms: Other symptoms such as swelling, restricted range of motion and mechanical symptoms; (3) KOOS ADL: Disability on the level of daily activities; (4) KOOS Sport/Rec: Disability on a level physically more demanding than activities of daily living; (5) KOOS QOL: Quality of life, mental and social aspects such as awareness and lifestyle changes. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Intermittent and Constant Osteoarthritis Pain (ICOAP) | 18 Months
  The ICOAP assesses pain in individuals with knee osteoarthritis taking into account both constant and intermittent pain experiences. Individual items are scored from 0 to 4. Each subscale (intermittent pain; constant pain; and total pain) are averaged. Lower numbers indicate lower pain.
Health Literacy | 18 Months
  Behavioral Risk Factor Surveillance System measures health literacy. Lower scores indicate higher literacy.
Cognitive Functioning | 18 Months
  The MOCA will be used to measure cognitive function. Scores range 0-30. Higher scores indicate higher cognitive functioning.
Brief Resilience Scale | 18 Months
  The Brief Resilience Scale will be used to measure resilience. The brief resilience scale (BRS) contains 6 items. The BRS is scored by reverse coding negatively worded questions (2, 4, and 6) and finding the mean of the six items. Range= 1-5. Lower scores indicate less resilience.
Physical Activity | 18 Months
  Physical activity will be measured by The Physical Activity Scale for the Elderly (PASE). 1-6 are scored in terms of hours per day over a 7-day period. Items 7-12 are scored as 1= engaged in activity or 0=did not engage in activity during the previous seven days. Scores range 0-100. Higher scores indicate more activity.
Depression - Center for Epidemiologic Studies Depression Scale (CES-D) | 18 Months
  Depression will be measured using the Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D contains 20-items and measures how often over the past week persons experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Health Related Quality of Life: Euroqol | 18 Months
  Compare the effects of a 6-month weight-loss maintenance intervention grounded in social cognitive theory to a health education intervention on health-related quality of life. The EQ-5D comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Responses results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Messier, PhD, Principal Investigator — Wake Forest University; Leigh Callahan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - Johnston County - UNC Chapel Hill, Chapel Hill, North Carolina
  - Haywood County - Haywood Regional Medical Center, Clyde, North Carolina
  - Forsyth County - Wake Forest University/Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The investigators support data sharing and will comply with all NIH guidelines as outlined in the NIH Data Sharing Policy and Implementation Guidance document. The primary means of data sharing and dissemination will be through scientific publications and presentations. Ensuring patient privacy and confidentiality will be of primary importance in creating the files to be shared. All data files will be de-identified. De-identification procedures will meet HIPAA criteria detailed in the Code of Federal Regulations, Part 46, Section 164.514. The study team will create a link on our website that describes the data files. Documentation will also be provided along with the redacted data files. The documentation will include electronic versions of the protocol, data collection forms (with instructions for scoring, if needed), data dictionary, data code book, labels, and formats. Requests for data will be answered via completion of an online request form and data-sharing agreement.
Supporting Information: Study Protocol, ICF
Time Frame: All data will be released within three years of completing collection, even if planned papers have not been written or accepted.

DOCUMENTS (1):
  • Informed Consent Form (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT03832296/ICF_000.pdf